CLINICAL TRIAL: NCT00758394
Title: Clinical Study to Compare Dental Plaque Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0907-PLA-14-RR
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2008-11-19 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; fluorophosphate; Triclosan; Sodium Fluoride; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluoride - A (Placebo Comparator): Fluoride only toothpaste
  Interventions: Drug: Fluoride
- Total + Whitening toothpaste - B (Active Comparator): Triclosan/fluoride toothpaste
  Interventions: Drug: Triclosan/Fluoride
- Triclosan/fluoride/Amino Acid - C (Experimental): toothpaste containing amino acid #1
  Interventions: Drug: Triclosan/Fluoride
- Triclosan/fluoride/Cavistat -D (Experimental): toothpaste containing amino acid/bicarbonate
  Interventions: Drug: Triclosan/Fluoride

INTERVENTIONS:
Drug: Fluoride — Brush two times a day for 4 days.
  Other Names: monofluorophosphate
  Arms: Fluoride - A
Drug: Triclosan/Fluoride — Brush two times daily for 4 days
  Other Names: sodium fluoride; triclosan
  Arms: Total + Whitening toothpaste - B
Drug: Triclosan/Fluoride — Brush twice daily for 4 days
  Other Names: sodium fluoride; triclosan; amino acid
  Arms: Triclosan/fluoride/Amino Acid - C
Drug: Triclosan/Fluoride — Brush twice daily for 4 days
  Other Names: sodium fluoride; triclosan; amino acid/bicarbonate
  Arms: Triclosan/fluoride/Cavistat -D

SUMMARY:
This clinical study was to evaluate the control of dental plaque formation after toothbrushing for 4 days with each of the 4 study toothpastes.

DETAILED DESCRIPTION:
Evaluation of dental plaque control for two prototype toothpastes will be determined by comparison to two control toothpastes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers at least 18 - 53 years of age
* Good general health
* Must sign informed consent form
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures
* Moderate or advanced periodontal disease or heavy dental tartar (calculus).
* 2 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that are currently affecting salivary function
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this study.
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Presence of an orthodontic appliance which interferes with plaque scoring.
* History of allergy to common dentifrice ingredients.
* History of allergy to arginine (amino acid)
* History of allergy to bicarbonate
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, Principal Investigator
Locations (1):
- Bluestone Center for Clinical Research, NYU College of Dentistry, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Groups:
- Fluoride First: Fluoride first, triclosan/fluoride second,Arginine/fluoride third and Cavistat/fluoride last
- Triclosan/Fluoride First: Triclosan fluoride first, Triclosan/fluoride/Arginine second, Triclosan/fluoride/Cavistat third, fluoride last
- Triclosan/Fluoride/Arginine First: Triclosan/fluoride/Arginine first, Triclosan/fluoride/Cavistat second,fluoride third, triclosan/fluoride last
- Triclosan/Fluoride/Cavistat First: Triclosan/fluoride/Cavistat first, fluoride second,Triclosan/fluoride third, Triclosan/fluoride/Arginine last
Period: 1st Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 8 | 7 | 6 | 8
Completed | 8 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout After 1st Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 8 | 7 | 6 | 8
Completed | 8 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: 2nd Intervention Order
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 8 | 7 | 6 | 8
Completed | 8 | 6 | 6 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Washout After 2nd Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 8 | 6 | 6 | 8
Completed | 8 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: 3rd Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 8 | 6 | 6 | 8
Completed | 7 | 6 | 6 | 7
Not Completed | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Period: Washout After 3rd Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 4th Intervention
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluoride - A: Negative control
- Fluoride/Triclosan - B: Positive control comparator
- Triclosan/Fluoride/Arginine: toothpaste containing amino acid
- Triclosan/Fluoride/Cavistat: toothpaste containing bicarbonate
- Total: Total of all reporting groups
Arm/Group | Fluoride - A | Fluoride/Triclosan - B | Triclosan/Fluoride/Arginine | Triclosan/Fluoride/Cavistat | Total
Number analyzed (Participants) | 8 | 7 | 6 | 8 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 6 | 8 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.8) | 29.7 (8.7) | 36.4 (11.6) | 37.8 (5.0) | 33.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 4 | 23
  Male | 2 | 0 | 0 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 6 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Index
Description: plaque units measured on a scale between 0 to 5. 0 = No plaque; 5 = 2/3 of Tooth covered in plaque.
Time Frame: 4-Day
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride - A | Fluoride/Triclosan - B | Triclosan/Fluoride/Arginine | Triclosan/Fluoride/Cavistat
Number analyzed (Participants) | 7 | 6 | 6 | 7
Units on a scale | 3.12 (0.38) | 2.90 (0.36) | 2.92 (0.42) | 2.94 (0.42)
Statistical Analysis 1: Comparison: Fluoride - A vs Fluoride/Triclosan - B vs Triclosan/Fluoride/Arginine vs Triclosan/Fluoride/Cavistat; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA — Two way Anova general linear model (subject and treatment as factors). Multiple comparison completed to determine differences between groups

ADVERSE EVENTS:
Time Frame: 8 weeks (including all washout periods and four (4) study intervention periods of 4 days each).
Arm/Group | Fluoride First | Triclosan/Fluoride First | Triclosan/Fluoride/Arginine First | Triclosan/Fluoride/Cavistat First
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days